CLINICAL TRIAL: NCT01669122
Title: A Randomized, Cross-Over, Single Dose Pharmacokinetic Study of 4mg Nicotine Lozenges.
Brief Title: Pharmacokinetic Study of 4 mg Nicotine Lozenge.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RH01333
Record Dates: First submitted 2012-08-16; First posted 2012-08-20 (Estimated); Results first posted 2015-01-22 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2014-10

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Prototype 1 (Experimental): 4mg nicotine lozenge administered orally as a single dose treatment per subject
  Interventions: Drug: nicotine
- Prototype 2 (Experimental): 4mg nicotine lozenge administered orally as a single dose treatment per subject
  Interventions: Drug: nicotine
- Prototype 3 (Experimental): 4mg nicotine lozenge administered orally as a single dose treatment per subject
  Interventions: Drug: nicotine
- Reference Therapy (Active Comparator): 4mg nicotine lozenge (internationally marketed) to be administered orally as a single dose treatment per subject.
  Interventions: Drug: nicotine

INTERVENTIONS:
Drug: nicotine — 4 mg nicotine lozenge experimental

SUMMARY:
This is a randomized, single center, open label, single dose, four way crossover study in fasted healthy male subjects to compare the pharmacokinetics of nicotine following administration of 3 prototype 4mg nicotine lozenge to an internationally marketed 4mg nicotine lozenge. Blood samples will be drawn at pre-specified intervals for a total of 12 hours post dose in each treatment session and plasma samples analyzed for nicotine levels.

ELIGIBILITY:
Inclusion Criteria:

- smoked commercially-manufactured cigarettes daily for the preceding 12 months and routinely smokes first cigarette within 30mins of awakening.

Exclusion Criteria:

* inability to refrain from smoking during confinement period, smoking tobacco in any other form other than commercially manufactured cigarettes, subject has used chewing tobacco or other tobacco products other than commercially manufactured cigarettes within 7 days of dosing

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Lambda Therapeutic Research Ltd, Ahmedabad, Gujarat, India

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the clinical site.
Pre-assignment Details: A total of 102 participants were screened, of which only 40 were randomized into the study. Fourteen participants did not meet the study criteria, 32 were lost to follow up, 2 withdrew consent while remaining 14 were not randomized due to other reasons.
Period: Period I
Arm/Group | Total Participants
Started | 40 (Participants who received Lozenge A=10, Lozenge B=10, Lozenge C=10, Reference Lozenge=10)
Safety Population | 39
Completed | 39
Not Completed | 1
Not completed — Lost to Follow-up | 1
Period: Washout Period I
Arm/Group | Total Participants
Started | 39
Completed | 39
Not Completed | 0
Period: Period II
Arm/Group | Total Participants
Started | 39 (Participants who received Lozenge A=9, Lozenge B=10, Lozenge C=10, Reference Lozenge=10)
Completed | 39
Not Completed | 0
Period: Washout Period II
Arm/Group | Total Participants
Started | 39
Completed | 37
Not Completed | 2
Not completed — Protocol Violation | 2
Period: Washout Period III
Arm/Group | Total Participants
Started | 37
Completed | 37
Not Completed | 0
Period: Period III
Arm/Group | Total Participants
Started | 37 (Participants who received Lozenge A=10, Lozenge B=8, Lozenge C=10, Reference Lozenge=9)
Completed | 37
Not Completed | 0
Period: Period IV
Arm/Group | Total Participants
Started | 37 (Participants who received Lozenge A=9, Lozenge B=10, Lozenge C=9, Reference Lozenge=9)
Completed | 37
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Safety Population: Baseline measurements were performed for safety population which included all participants in the study who were dispensed at least one of the study treatment. Out of 40 randomized participants, one participant did not receive any treatment and was lost to follow-up.
Arm/Group | Safety Population
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.7 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 39

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time 0 to t, AUC (0-t)
Description: Area under the plasma concentration time curve from zero and extrapolated to the time of last quantifiable sample was determined from plasma concentration time profile of nicotine. AUC(0 -t) was based on the baseline adjusted nicotine plasma concentration data.
Time Frame: Blood samples were collected pre-dose and at 5, 10, 15, 30 and 45 minutes and 1, 1.5, 2, 3, 4, 6, 8, 10 and 12 hours post dosing
Population: Per protocol (PP) population: all randomized participants profiles, without a protocol deviation that would have lead to the data exclusion.
Measure: Mean (Standard Deviation); unit: nanograms (ng)*hours (h)/milliliter (mL)
Groups:
- Test Lozenge (A): 4 mg nicotine lozenge with excipient A, was administered orally as a single dose treatment.
- Test Lozenge (B): 4 mg nicotine lozenge with excipient B, was administered orally as a single dose treatment.
- Test Lozenge (C): 4 mg nicotine lozenge with excipient C, was administered orally as a single dose treatment.
- Reference Lozenge: Reference 4 mg nicotine lozenge, was administered orally as a single dose treatment.
Arm/Group | Test Lozenge (A) | Test Lozenge (B) | Test Lozenge (C) | Reference Lozenge
Number analyzed (Participants) | 38 | 37 | 39 | 38
nanograms (ng)*hours (h)/milliliter (mL) | 89.14 (44.777) | 87.38 (42.816) | 86.60 (36.191) | 91.97 (45.601)
Statistical Analysis 1: Comparison: Test Lozenge (A) vs Reference Lozenge; Null hypothesis considered no difference in the treatments being compared; Test type: Non-Inferiority or Equivalence — Testing Bioequivalence; Treatment Ratio = 0.96, 90% CI 2-sided [0.93 to 0.99]
Statistical Analysis 2: Comparison: Test Lozenge (B) vs Reference Lozenge; Null hypothesis considered no difference in the treatments being compared; Test type: Non-Inferiority or Equivalence — Testing Bioequivalence; Treatment Ratio = 0.96, 90% CI 2-sided [0.93 to 0.99]
Statistical Analysis 3: Comparison: Test Lozenge (C) vs Reference Lozenge; Null hypothesis considered no difference in the treatments being compared; Test type: Non-Inferiority or Equivalence — Testing Bioequivalence; Treatment Ratio = 0.94, 90% CI 2-sided [0.91 to 0.97]

2. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: Maximum plasma nicotine concentration was determined from plasma-concentration time profiles. Cmax was based on the baseline adjusted nicotine plasma concentration data.
Time Frame: as for outcome 1
Population: PP population: all randomized participants profiles, without a protocol deviation that would have lead to the data exclusion.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Test Lozenge (A): 4 mg nicotine lozenge with excipient A was administered orally as a single dose treatment.
Arm/Group | Test Lozenge (A) | Test Lozenge (B) | Test Lozenge (C) | Reference Lozenge
Number analyzed (Participants) | 38 | 37 | 39 | 38
ng/mL | 18.50 (5.626) | 18.39 (5.099) | 17.41 (4.796) | 18.97 (6.001)
Statistical Analysis 1: Comparison: Test Lozenge (A) vs Reference Lozenge; Null hypothesis considered no difference in the treatments being compared; Test type: Non-Inferiority or Equivalence — Testing bioequivalence; Treatment Ratio = 0.97, 90% CI 2-sided [0.93 to 1.02]
Statistical Analysis 2: Comparison: Test Lozenge (B) vs Reference Lozenge; Null hypothesis considered no difference in the treatments being compared; Test type: Non-Inferiority or Equivalence — Testing Bioequivalence; Treatment Ratio = 0.99, 90% CI 2-sided [0.94 to 1.03]
Statistical Analysis 3: Comparison: Test Lozenge (C) vs Reference Lozenge; Null hypothesis considered no difference in the treatments being compared; Test type: Non-Inferiority or Equivalence — Testing Bioequivalence; Treatment Ratio = 0.92, 90% CI 2-sided [0.88 to 0.96]

3. Secondary Outcome: AUC(0-inf)
Description: Area under the plasma nicotine concentration-time curve from zero extrapolated to infinity was determined. AUC(0-inf) was based on the baseline adjusted nicotine plasma concentration data.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Test Lozenge (A) | Test Lozenge (B) | Test Lozenge (C) | Reference Lozenge
Number analyzed (Participants) | 38 | 37 | 39 | 38
ng*hr/mL | 100.33 (60.132) | 98.90 (61.958) | 97.83 (52.324) | 104.53 (65.525)
Statistical Analysis 1: Comparison: Test Lozenge (A) vs Reference Lozenge; Null hypothesis considered no difference in the treatments being compared; Test type: Non-Inferiority or Equivalence — Testing bioequivalence; Treatment Ratio = 0.96, 90% CI 2-sided [0.93 to 0.99]
Statistical Analysis 2: Comparison: Test Lozenge (B) vs Reference Lozenge; Null hypothesis considered no difference in the treatments being compared; Test type: Non-Inferiority or Equivalence — Testing bioequivalence; Treatment Ratio = 0.96, 90% CI 2-sided [0.93 to 0.99]
Statistical Analysis 3: Comparison: Test Lozenge (C) vs Reference Lozenge; Null hypothesis considered no difference in the treatments being compared; Test type: Non-Inferiority or Equivalence — Testing bioequivalence; Treatment Ratio = 0.93, 90% CI 2-sided [0.90 to 0.96]

4. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax)
Description: Tmax was determined from plasma concentration time profiles. Tmax was based on the baseline adjusted nicotine plasma concentration data.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Test Lozenge (A) | Test Lozenge (B) | Test Lozenge (C) | Reference Lozenge
Number analyzed (Participants) | 38 | 37 | 39 | 38
hours | 1.50 [0.50 to 4.00] | 1.50 [0.25 to 6.00] | 1.50 [0.75 to 6.00] | 1.50 [0.25 to 3.00]
Statistical Analysis 1: Comparison: Test Lozenge (A) vs Reference Lozenge; Null hypothesis considered no difference in the treatments being compared; Test type: Superiority or Other; p = 0.2208, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.00, 95% CI 2-sided [0.00 to 0.50] — Based on Hodges Lehmann estimate
Statistical Analysis 2: Comparison: Test Lozenge (B) vs Reference Lozenge; Null hypothesis considered no difference in the treatments being compared; Test type: Superiority or Other; p = 0.5695, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.00, 95% CI 2-sided [-0.25 to 0.25] — Based on Hodges Lehmann estimate
Statistical Analysis 3: Comparison: Test Lozenge (C) vs Reference Lozenge; Null hypothesis considered no difference in the treatments being compared; Test type: Superiority or Other; p = 0.0063, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.00, 95% CI 2-sided [0.00 to 0.50] — Based on Hodges Lehmann estimate

5. Secondary Outcome: Rate of Elimination (Kel)
Description: Elimination rate constant for nicotine was calculated. Kel was based on the baseline adjusted nicotine plasma concentration data.
Time Frame: Blood samples were collected pre-dose at 5, 10, 15, 30 and 45 minutes and 1, 1.5, 2, 3, 4, 6, 8, 10 and 12 hours post dosing
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 1/ hour
Arm/Group | Test Lozenge (A) | Test Lozenge (B) | Test Lozenge (C) | Reference Lozenge
Number analyzed (Participants) | 38 | 37 | 39 | 38
1/ hour | 0.26 (0.06) | 0.26 (0.07) | 0.27 (0.11) | 0.26 (0.07)

6. Secondary Outcome: Plasma Half Life (t1/2)
Description: Half-life of elimination of nicotine was determined. t1/2 was based on the baseline adjusted nicotine plasma concentration data.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Test Lozenge (A) | Test Lozenge (B) | Test Lozenge (C) | Reference Lozenge
Number analyzed (Participants) | 38 | 37 | 39 | 38
hours | 2.86 (0.80) | 2.91 (0.99) | 2.86 (1.07) | 2.94 (0.99)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the start of the treatment, and until 7 days following administration of the last dose of investigational product.
Arm/Group | Test Lozenge (A) | Test Lozenge (B) | Test Lozenge (C) | Reference Lozenge
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/37 | 0/39 | 0/38
Other Adverse Events (participants affected / at risk) | 0/38 | 0/37 | 0/39 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.